CLINICAL TRIAL: NCT01697761
Title: Efficacy of Acupuncture and Moxibustion Treatment in Patients With Active Crohn's Disease and Its Regulation Mechanism to the Immune Homeostasis Mediated by Th17/Treg Cells
Brief Title: Efficacy of Acupuncture and Moxibustion Treatment in Patients With Active Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHACU-201202
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2012-09

CONDITIONS: Crohn's Disease; CAM
Keywords: Crohn's disease,acupuncture,moxibustion,inflammation factors
MeSH Terms: conditions — Crohn Disease | interventions — Acupuncture Therapy; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): treat by moxibustion and acupuncture
  Interventions: Other: Treatment Group
- Control Group (Experimental): treat by Sham acupuncture and moxibustion
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Treatment Group — patients receive herbs-partitioned moxibustion for 2 cones and acupuncture for 30 minutes，3 times a week for 12 weeks
  Other Names: acupuncture and moxibustion group; acupuncture and Herbs-partitioned moxibustion group
  Arms: Treatment Group
Other: Control Group — patients receive shallow needing and bran-partitioned moxibustion with the stimulation same to the treatment group.
  Other Names: Sham acupuncture and moxibustion group
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether acupuncture or moxibustion therapies are effective in the treatment of active Crohn's disease. meanwhile, we are aim to observe the content of Inflammatory factors and Neurotransmitter before and after acupuncture and moxibustion therapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether acupuncture or moxibustion therapies are effective in the treatment of active Crohn's disease. meanwhile, we are aim to observe the content of Inflammatory factors and Neurotransmitter before and after acupuncture and moxibustion therapy.

Through treating active Crohn's disease by acupuncture and moxibustion therapies for 12 weeks, we are aim to observe the efficiency and the probably change of Inflammatory factors and Neurotransmitter of colonic mucosa and we may elucidate the mechanism of the efficiency of acupuncture and moxibustion therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years;
* Crohn's Disease Activity Index [CDAI]>150 and <450;
* not taking any medication or taking salicylates, prednisone ( dose≤ 15mg and at least have taken a month ), after entering the study the dose remained constant;
* Not taking immunosuppressive agents or use " with " biological preparations within 3 months prior to entering the study
* signing a written informed consent form.

Exclusion Criteria:

* Severe Crohn's disease patients or patients in remission ( CDAI > 450 or < 150 );
* The pregnancy or lactation period patients ;
* patients associated with heart, brain, liver, kidney and hematopoietic system disease;
* The psychiatric patients;
* Patients with other serious diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
CDAI | 2 years
  Crohn's Disease Activity Index

SECONDARY OUTCOMES:
Inflammatory factors | 2 years
  Intestinal mucosa of Th17/Treg,IL-6,IL-17,IL-23,etc
Neurotransmitter | 2 years
  Intestinal mucosa of 5-HT,DA,SP,VIP and their receptors etc
IBDQ | 2 years
  Inflammatory Bowel Disease Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wu Huangan, PhD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian
Locations (1):
- Shanghai Institute of Acupuncture-Moxibustion and Merdian, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Bao CH, Zhao JM, Liu HR, Lu Y, Zhu YF, Shi Y, Weng ZJ, Feng H, Guan X, Li J, Chen WF, Wu LY, Jin XM, Dou CZ, Wu HG. Randomized controlled trial: moxibustion and acupuncture for the treatment of Crohn's disease. World J Gastroenterol. 2014 Aug 21;20(31):11000-11. doi: 10.3748/wjg.v20.i31.11000. PMID 25152604